CLINICAL TRIAL: NCT03222388
Title: Electronic Validation of the International Index of Erectile Function Questionnaire (IIEF) 5 and 15.
Brief Title: Electronic IIEF Validation
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Société Internationale d'Urologie (Other)
Responsible Party: Principal Investigator, Prof.dr. J.J.M.C.H. de la Rosette, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 17.281
Record Dates: First submitted 2017-06-27; First posted 2017-07-19 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Erectile Dysfunction
Keywords: IIEF; electronic validation
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- IIEF5 paper-electronic
  Interventions: Other: Questionnaire - IIEF 5/15
- IIEF5 electronic-paper
  Interventions: Other: Questionnaire - IIEF 5/15
- IIEF15 paper-electronic
  Interventions: Other: Questionnaire - IIEF 5/15
- IIEF15 electronic-paper
  Interventions: Other: Questionnaire - IIEF 5/15
- IIEF5 electronic-electronic
  Interventions: Other: Questionnaire - IIEF 5/15
- IIEF15 electronic-electronic
  Interventions: Other: Questionnaire - IIEF 5/15

INTERVENTIONS:
Other: Questionnaire - IIEF 5/15 — International Index of Erectile Function

SUMMARY:
Questionnaires are used within urology to objectify disease burden and symptom changes during therapy. Recent technological improvements, as the smartphone and tablet, create new fill-out possibilities. However, questionnaires are only validated on paper. In order to use questionnaires for multiple platforms, electronic validation is needed. The International Prostate Symptom Score has already been validated on the smartphone. The International Index of Erectile Function (normal version of 15 questions and short version of 5 questions) is widely used within urology, however electronic validation is required for usage on electronic platforms in the future.

ELIGIBILITY:
Inclusion criteria:

* Male patients, ≥40 years of age, presenting at the outpatient clinic of Urology of the Academic Medical Center in Amsterdam.
* In possession of a smartphone, tablet or laptop/computer with internet connection.
* Access to email.
* Fluent speaking and reading the Dutch language.

Exclusion criteria:

* Change in treatment, especially erectile dysfunction at consultation which could impact the short term IIEF outcome during the cross-over time.
* Unable to provide informed consent.
* Unfit according to the medical doctor (for example cognitive problems, leading to inadequate follow-up of instructions).

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be included at the outpatient clinic of the urology department at the Academic Medical Center in Amsterdam.
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Reliability | Per subject, thus 7 days.
  The electronic IIEF-5 and 15 questionnaire is reliable when the ICC is ≥0.7, when compared with the paper version.

SECONDARY OUTCOMES:
Preference for paper or electronic | Per subject, after 7 days.
  The electronic version of the IIEF-5 and 15 is preferred when ≥70% of the subjects have no preference or prefer the electronic version over the paper version.

CONTACTS AND LOCATIONS:
Locations (1):
- AMC University Hospital, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Kollenburg RAA, de Bruin DM, Wijkstra H. Validation of the Electronic Version of the International Index of Erectile Function (IIEF-5 and IIEF-15): A Crossover Study. J Med Internet Res. 2019 Jul 2;21(7):e13490. doi: 10.2196/13490. PMID 31267983